CLINICAL TRIAL: NCT00109564
Title: A Safety and Efficacy Study of TC-1734-112 in Subjects With Age Associated Memory Impairment (AAMI)
Brief Title: A Safety and Efficacy Study of Ispronicline (TC-1734-112) in Subjects With Age Associated Memory Impairment (AAMI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TC-1734-112-CRD-004
Record Dates: First submitted 2005-04-28; First posted 2005-04-29 (Estimated); Last update posted 2008-07-18 (Estimated); Status verified 2008-07

CONDITIONS: Age-Related Memory Disorders
Keywords: AAMI; Memory Impairment; Decline in Cognitive Function; Age Associated Memory Impairment
MeSH Terms: conditions — Memory Disorders | interventions — ispronicline; Nicotinic Agonists

INTERVENTIONS:
Drug: ispronicline (nicotinic acetylcholine receptor agonist)

SUMMARY:
The purpose of this Phase II study is to evaluate the efficacy and safety of ispronicline (TC-1734-112) compared to placebo (inactive substance pill) in patients with age associated memory impairment (AAMI). AAMI is characterized as cognitive impairment including memory loss and poor concentration associated with aging.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 50-80 years.
* Lives with a significant other.
* Has subjective memory complaints. Verbal verification of this subjective memory complaint will be obtained from the significant other.
* Has no severe, uncontrolled medical condition.
* If receiving treatment for a medical condition, that treatment has been stable for at least 2 months before entering the trial and to remain stable throughout the trial.

Exclusion Criteria

* Aged less than 50 years or greater than 80 years.
* Lives alone.
* Has any medical condition not adequately controlled, or likely to interfere with performance of the study procedures.
* Medication for a medical condition has been changed in the last 2 months or during the trial.
* Administration of acetylcholinesterase inhibitors and gingko biloba within 2 months prior to entering the study.
* Has evidence of depression or anxiety
* Meets DSM-IV criteria for Alzheimer's or vascular dementia.
* Has participated in an investigational drug trial in the previous 30 days.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174
Dates: Start 2005-01; Study Completion 2005-10

PRIMARY OUTCOMES:
To assess safety and tolerability of ispronicline vs. placebo in generally healthy elderly subjects with subjective and objective memory impairment meeting the generally accepted criteria for AAMI.
To assess effect, on cognition, of ispronicline vs. placebo in generally healthy elderly subjects with subjective and objective memory impairment meeting the generally accepted criteria for AAMI.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Pivotal Research Center, Mesa, Arizona
  - Pivotal Research Center, Peoria, Arizona
  - Radiant Research, Denver, Colorado
  - Neuropsychiatric Research Center of SW Florida, Fort Meyers, Florida
  - Meridien Research, Saint Petersberg, Florida
  - Meridien Research, Tampa, Florida
  - Northlake Medical Research Center, Decatur, Georgia
  - Hartford Research, Florence, Kentucky
  - Berman Center, Minneapolis, Minnesota
  - Radiant Research, St Louis, Missouri
  - Kulynych Research Center, Greensboro, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Radiant Research Philadelphia, Philadelphia, Pennsylvania
  - Radiant Research, San Antonio, Texas
  - Radiant Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Dunbar GC, Kuchibhatla RV, Lee G; TC-1734 (AZD3480) AAMI Clinical Study Group (USA). A randomized double-blind study comparing 25 and 50 mg TC-1734 (AZD3480) with placebo, in older subjects with age-associated memory impairment. J Psychopharmacol. 2011 Aug;25(8):1020-9. doi: 10.1177/0269881110367727. Epub 2010 Jun 11. PMID 20542923